CLINICAL TRIAL: NCT00052104
Title: A Telephone Intervention for Dementia Caregivers
Brief Title: Telephone-Based Support for Caregivers of Patients With Dementia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21MH062561 (NIH); R21MH062561 (NIH); DSIR GT-GS
Record Dates: First submitted 2003-01-22; First posted 2003-01-23 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2008-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Family Systems Intervention

SUMMARY:
The purpose of this study is to develop an effective, low-cost, telephone-based intervention to reduce anxiety, depression, and feelings of burden and stress in caregivers of patients with dementia. This study will also determine whether the intervention can alter the course of dementia.

DETAILED DESCRIPTION:
Caregivers are randomized to receive either telephone-based intervention or standard medical care. Both groups receive a resource packet containing information about caring for someone with dementia and a list of local resources. Caregivers in the intervention group also receive a series of telephone calls over 12 months, during which education, emotional support, and training in problem-solving skills are provided by trained therapists. Caregivers in the standard care group receive no additional psychosocial intervention. Participants are assessed pre-treatment, mid-treatment (6 months), post-treatment, and at a 3-month follow-up.

ELIGIBILITY:
Patient Inclusion Criteria:

* DSM-IV diagnosis of dementia (vascular, mixed, or associated with Alzheimer's disease)
* Lives in the community, including senior/retirement centers, but excluding nursing homes and assisted living centers
* 50 years old or older
* Resides in Southeastern New England

Caregiver Inclusion Criteria:

* Living with a person with dementia
* Provides care for at least 6 months for at least 4 hours a day
* English as primary language
* Telephone access
* Resides in Southeastern New England

Patient Exclusion Criteria:

* Major acute medical condition affecting independent functioning

Caregiver Exclusion Criteria:

* Acute medical illness
* Cognitive impairment as defined by an MMSE score < 25

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2001-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States